CLINICAL TRIAL: NCT04074096
Title: Randomised Phase 2 Trial Testing the Addition of Upfront Stereotactic Radiosurgery to Binimetinib Encorafenib Pembrolizumab Compared to Binimetinib Encorafenib Pembrolizumab Alone in BRAFV600 Mutation-positive Melanoma With Brain Metastasis
Brief Title: Binimetinib Encorafenib Pembrolizumab +/- Stereotactic Radiosurgery in BRAFV600 Melanoma With Brain Metastasis
Acronym: BEPCOME-MB
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: European Association of Dermato Oncology (Unknown); Pierre Fabre Medicament (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD06 - UC-0107/1810; 2021-006331-26 (EudraCT Number)
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Malignant Melanoma; BRAF V600 Mutation; Brain Metastases
Keywords: Melanoma; BRAF V600; Brain metastases; Encorafenib; Binimetinib; Pembrolizumab; Stereotaxic; SRS
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Radiosurgery; binimetinib; encorafenib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encorafenib + binimetinib + pembrolizumab (Experimental): Encorafenib 450 mg oral route (PO) once daily (QD) + binimetinib 45 mg PO twice daily (BID) + pembrolizumab 200 mg intravenous (IV) every 3 weeks (Q3W).
  Interventions: Drug: Binimetinib Oral Tablet; Drug: Encorafenib Oral Capsule; Drug: Pembrolizumab
- SRS followed by encorafenib + binimetinib + pembrolizumab (Experimental): Upfront SRS of all lesions ≥5 mm in diameter (or ≥3 mm if other cerebral metastases >5 mm); followed by encorafenib 450 mg PO QD + binimetinib 45 mg PO BID + pembrolizumab 200 mg IV Q3W. The treatment should be started more than 24 hours and less than 8 days (excluded) after the SRS
  Interventions: Radiation: Stereotaxic radiosurgery (SRS); Drug: Binimetinib Oral Tablet; Drug: Encorafenib Oral Capsule; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotaxic radiosurgery (SRS) — For patients randomised to arm B only: Upfront SRS of all lesions ≥5 mm in diameter (or ≥3 mm if other cerebral metastases >5 mm).
  Arms: SRS followed by encorafenib + binimetinib + pembrolizumab
Drug: Binimetinib Oral Tablet — All patients: binimetinib 45 mg PO BID.
  Other Names: Mektovi
Drug: Encorafenib Oral Capsule — All patients: encorafenib 450 mg PO QD
  Other Names: Braftovi
Drug: Pembrolizumab — All patients: pembrolizumab 200 mg IV Q3W
  Other Names: Keytruda

SUMMARY:
This study evaluates the addition of stereotactic radiosurgery (SRS) to the combination of binimetinib + encorafenib + pembrolizumab in the treatment of BRAFⱽ⁶⁰⁰ mutation-positive melanoma with brain metastases (MBM).

DETAILED DESCRIPTION:
This is a Phase 2, randomised, controlled, open-label, multicentric, parallel trial with a safety lead-in phase, to assess the efficacy and safety of adding upfront SRS to binimetinib-encorafenib-pembrolizumab combination therapy in the treatment of BRAFⱽ⁶⁰⁰ mutation-positive MBM.

The study will incorporate a safety lead-in (SLI) phase to assess the tolerability of binimetinib-encorafenib-pembrolizumab combination therapy +/- SRS in the first six patients enrolled. Safety will be assessed by the occurrence of predefined dose limiting toxicity (DLT) events. The safety data will be reviewed by an independent data monitoring committee (IDMC).

The trial plans to enrol 150 patients who will be randomly assigned (1:1) to receive treatment with either:

* Arm A: Encorafenib + binimetinib + pembrolizumab
* Arm B: Upfront stereotactic radiosurgery of all lesions ≥5 mm in diameter (or ≥3 mm if other cerebral metastases >5 mm); followed by encorafenib + binimetinib + pembrolizumab . The treatment should be started more than 24 hours and less than 8 days (excluded) after the SRS.

Patients will be treated until disease progression. Pembrolizumab will be discontinued after a maximum of 35 administrations. Treatment may also be terminated early at the initiative of either the patient or the investigator for any reason that would be beneficial to the patient

All patients will be followed for a total of 5 years post-randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent prior to any trial specific procedures.
2. Aged ≥18 years old.
3. An Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
4. Histologically confirmed Stage IV M1d cutaneous melanoma or unknown primary melanoma that is metastatic to the brain.
5. Presence of BRAFV600E/K/D/R mutation according to a locally validated BRAF Assay.
6. Candidacy for SRS therapy validated by the radiation oncologist and/or neurosurgeon at the investigative centre. This should be documented in the patient file.
7. Absence of previous systemic treatment with BRAF inhibitors, MEK inhibitors or anti-PD-1 for distant metastatic melanoma. Patients having received such treatments as adjuvant therapy are allowed provided adjuvant treatment has been stopped for 6 months or more.
8. No more than one previous local intracranial therapy for one lesion (e.g. craniotomy, SRS).

   Note: Treatment with stereotactic radiosurgery must have been completed ≥14 days prior to randomisation and this lesion cannot be target lesion for radiosurgery.
9. Able to undergo gadolinium-enhanced MRI.
10. At least one measurable intracranial lesion for which all of the following criteria have to be met:

    1. Previously untreated (no local therapy including local radiotherapy, resection, radiosurgery) or progressive after previous local therapy.
    2. Longest diameter ≥5 mm as determined by contrast-enhanced MRI. Longest diameter ≥3 mm is acceptable for other IC lesions provided there is at least one lesion ≥5 mm.
    3. Cumulative Intracranial Target Volume ≤12 cmᵌ as determined by contrast-enhanced MRI.
11. All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values) must be resolved or Grade 1 according to NCI-CTCAE v5.0.
12. Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption (malabsorption syndrome, major resection of the stomach or bowels).
13. Adequate bone marrow, organ function, and laboratory parameters defined as the following (all criteria must be met):

    1. Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L;
    2. Haemoglobin ≥9 g/dL without transfusions;
    3. Platelets ≥100 x 10⁹/L without transfusions;
    4. Aspartate aminotransferase and alanine aminotransferase ≤2.5 × upper limit of normal (ULN); ≤5 x ULN is acceptable for patient with liver metastases;
    5. Total bilirubin ≤2 x ULN;
    6. Creatinine ≤1.5 mg/dL, or calculated creatinine clearance ≥50 mL/min (as determined using the MDRD method).
14. Adequate cardiac function, defined as the following (all criteria must be met):

    * Left ventricular ejection fraction (LVEF) ≥ local lower normal limit (LLN) as determined by a multigated acquisition (MUGA) scan or echocardiogram;
    * Baseline QT interval corrected for heart rate QTc ≤ 480 ms according to local standard formula.
15. Women of childbearing potential (WOCBP) or men must agree to refrain from sexual activity or use adequate contraception for the duration of study treatment and for 120 days after completing treatment. Male participants must agree to refrain from donating sperm during this period.
16. Patient affiliated to or a beneficiary of the local social security system or equivalent.
17. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

1. More than 10 intracranial metastases.
2. Presence of neurological symptoms related to intracranial metastases which induce alteration of the ECOG performance status to 2 or more or require immediate radiation treatment.
3. Ocular melanoma.
4. Brain metastases which necessitate immediate neurosurgery.
5. Any previous treatment with whole-brain radiation.
6. Presence of leptomeningeal disease or any parenchymal brain metastasis >30 mm in longest diameter.

   Note: On MRI, the most common finding of leptomeningeal disease is pial enhancement and nodularity, typically over the cerebral convexities, in the basal cisterns, on the tentorium, or in the ventricular ependymal surfaces.
7. Current or expected use of a strong inhibitor of CYP3A4.
8. History of malignancy other than disease under study occurring within 3 years of study enrolment with the exception of: completely resected non-melanoma skin cancer or indolent second malignancies.
9. Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that, in the opinion of the investigator, could interfere with the patient's safety, obtaining informed consent, or compliance with study procedures.
10. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (patients with laboratory evidence of cured HBV and/or HCV will be permitted).
11. A history or evidence of cardiovascular risk including any of the following:

    1. Left ventricular ejection fraction < local LLN as determined by a MUGA scan or echocardiogram;
    2. A QT interval corrected for heart rate QTc > 480 ms according to local standard formula;
    3. A history or evidence of current clinically significant uncontrolled arrhythmias.

       Note: Patients with atrial fibrillation controlled for >30 days prior to randomisation are eligible.
    4. A history or evidence of current >Class II congestive heart failure as defined by the New York Heart Association guidelines;
    5. Treatment refractory hypertension defined as a systolic blood pressure of >140 mmHg and/or diastolic blood pressure >90 mmHg, which cannot be controlled by antihypertensive therapy;
    6. Patients with intra-cardiac defibrillators;
    7. A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting less than 6 months prior to enrolment.
12. A history or current evidence of retinal vein occlusion.
13. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, and their excipients.
14. Hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
15. Participation in another therapeutic trial within the 30 days prior to randomization
16. Pregnant or breastfeeding female. Note: WOCBP must have a negative serum pregnancy test within 14 days prior to enrolment.
17. History of, or active interstitial lung disease or (non-infectious) pneumonitis.
18. Active, known or suspected autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease (Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll).
19. Diagnosis of immunodeficiency or systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date for first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.
20. Has received a live vaccine within 30 days prior to the first dose of study drug.
21. Active infection requiring systemic therapy.
22. Known history of active TB (Bacillus Tuberculosis).
23. Allogenic tissue/solid organ transplant.
24. Person deprived of their liberty or under protective custody or guardianship.
25. Patient unwilling or unable to comply with the medical follow-up required by the trial because of geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Intracranial (IC) progression-free survival (PFS) | From randomisation until IC-PD, or death, whichever occurs first, up to 12 months.
  Time from randomisation until IC-progressive disease (PD) as evaluated by centralized assessment using modified response evaluation criteria in solid tumours version 1.1 (RECIST v1.1), or death, whichever occurs first.

SECONDARY OUTCOMES:
Intracranial-response rate (RR) | From randomisation until IC-CR or IC-PR, up to 60 months.
  Percentage of patients with a confirmed IC-complete response (CR) or IC-partial response (PR) as assessed by the investigator using modified RECIST v1.1.
Intracranial disease control (DC) | From randomisation until IC-CR or IC-PR or stable intracranial disease, up to 60 months.
  Percentage of patients with an IC-CR or IC-PR or stable intracranial disease as assessed by the investigator using modified RECIST v1.1.
Extracranial (EC) response rate | From randomisation until confirmed EC-CR or EC-PR, up to 60 months.
  Percentage of patients with a confirmed EC-CR or EC-PR as assessed by the investigator using modified RECIST v1.1.
Overall response rate (ORR) | From randomisation until confirmed CR or PR, up to 60 months.
  Percentage of patients with a confirmed CR or PR as assessed by the investigator using modified RECIST v1.1 to assess IC-response and RECIST v1.1 for EC-response.
Duration of intracranial, extracranial, and overall response | Time from first observation of, IC-, EC-, or overall response respectively (i.e. CR or PR), until disease progression (PD), up to 60 months.
  Time from first observation of, IC-, EC-, or overall response respectively (i.e. CR or PR), until disease progression (PD) according to modified RECIST v1.1 (intracranial disease) or RECIST v1.1 (extracranial disease) or death, whichever occurs first.
Duration of response of treated target lesions | From first documented response (i.e. CR or PR) until PD of treated target lesions or death, whichever occurs first, up to 60 months.
  Time from first documented response (i.e. CR or PR) until PD of treated target lesions or death, whichever occurs first.
Progression-free survival (PFS) | From randomisation until IC-PD, EC-PD or death, whichever occurs first, up to 60 months.
  Time from randomisation until IC-PD according to modified RECIST v1.1, EC-PD according to RECIST v1.1, or death, whichever occurs first.
Overall survival (OS) | From randomisation until death due to any cause, up to 60 months.
  Time from randomisation until death due to any cause.
Global Quality of Life (HRQOL) - QLQ-C30 | From randomisation until end of treatment, up to 60 months.
  This self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life (HRQOL) in patients with brain metastases - QLQ-BN20 | From randomisation until end of treatment, up to 60 months.
  This EORTC brain cancer specific questionnaire is intended to supplement the QLQ-C30 questionaire.
  The QLQ-BN20 contains 20 items organized into four scales (three items each: future uncertainty, visual disorder, motor dysfunction, and communication deficit), and seven single items (headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs, and bladder control). All items are rated on a four-point Likert-type scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Cognitive performance | From randomisation until end of treatment, up to 60 months.
  Assessed using the Montreal Cognitive Assessment (MoCA).
Incidence of dose-limiting toxicities | From randomisation until completion of 2 cycles of treatment
  Occurrence of adverse events predefined as dose-limiting toxicities in any patient during the safety lead-in phase of the trial
Frequency and severity of adverse events | From randomisation until end of treatment, up to 60 months.
  Assessed according to National Cancer Institute - Common terminology criteria for adverse events version 5.0 (NCI-CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Saiag, Prof, Principal Investigator — APHP - CHU Ambroise Paré; Marie Charissoux, MD, Principal Investigator — Institut Régional du Cancer; Jean Regis, Prof, Principal Investigator — APHM - Hôpital de la Timone
Locations (21):
- France (21):
  - APHP - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux
  - GH Sud CHU Bordeaux - Hôpital Levêque, Bordeaux
  - APHP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Caen, Caen
  - CLCC - Centre Jean François Baclesse, Caen
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hopital Du Bocage, Dijon
  - CLCC - Centre Georges François Leclerc, Dijon
  - CLCC - Centre Léon Bérard, Lyon
  - APHM - Hopital De La Timone, Marseille
  - CHU De Montpellier - Hopital Saint Eloi, Montpellier
  - CLCC - Institut de Cancerologie de Montpellier, Montpellier
  - CHU Nice - Hôpital de l'Archet, Nice
  - CLCC - Centre Antoine Lacassagne, Nice
  - APHP - L'hôpital de la Pitié-Salpêtrière, Paris
  - CHU de Nantes - Hôtel Dieu, Saint-Herblain
  - CLCC - Institut de Cancerologie de l'Ouest - Nantes, Saint-Herblain
  - CLCC - IUCT-0 / Institut Claudius Regaud, Toulouse
  - CHU de TOURS - Hôpital Bretonneau, Tours
  - CLCC - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.